CLINICAL TRIAL: NCT06262269
Title: Interest of Adapted Physical Activity by Tele-rehabilitation in Chronic Pathology - Application to Idiopathic Scoliosis in Adolescents
Brief Title: Interest of Adapted Physical Activity by Tele-rehabilitation in Chronic Pathology - Idiopathic Scoliosis in Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Association des Paralysees de France (APF) (Other)
Collaborators: Fondation de France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sportscol; 2022-A00021-42 (Other: Number IDRCB)
Record Dates: First submitted 2023-02-01; First posted 2024-02-16 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: Adapted physical activity; Telerehabilitation; Physical condition; Hiit; Exercise booklet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TELE-APA (Experimental): The TELE-APA group will benefit from an individual, specific HIIT type program, adapted to the scoliosis of each patient, by tele-rehabilitation, supervised by a teacher in adapted physical activities during 12 weeks. Then he will benefit from an adapted physical activity program at home, based on a booklet of specific exercises identical to that of the CONTROL group, of HIIT type, adapted to the scoliosis of adapted to the scoliosis of each patient for 12 weeks.
  Interventions: Other: Home-based adapted physical activity program supervised by an APA teacher via individual video conference.; Other: Second period of the home-based adapted physical activity program with an exercise booklet.
- CONTROL (Active Comparator): The CONTROL group will benefit from an adapted physical activity program at home, based on a booklet of specific HIIT-type exercises, adapted to the scoliosis of each patient for 2 times 12 weeks. A new exercise booklet is given at the end of the first 12 weeks.
  Interventions: Other: First period of the home-based adapted physical activity program with an exercise booklet.; Other: Second period of the home-based adapted physical activity program with an exercise booklet.

INTERVENTIONS:
Other: Home-based adapted physical activity program supervised by an APA teacher via individual video conference. — Participants will follow a 12-week tele-rehabilitation programme involving high-intensity interval training (HIIT) adapted to their AIS. The programme includes three 45-minute individual sessions per week. The exercises are selected from a database designed for AIS patients. The APA teacher will systematically document the patient's presence or absence at each tele-rehabilitation session, thus assessing their adherence to the programme.
  Other Names: Period 1 - TELE-APA
  Arms: TELE-APA
Other: First period of the home-based adapted physical activity program with an exercise booklet. — Participants will receive a self-programme in the form of a booklet of specific HIIT-type exercises adapted to their AIS. The programme is to be carried out at home over a 12-week period, with 3 45-minute sessions per week. The exercises are taken from the same database. Each participant in the CONTROL group will be encouraged to keep a follow-up diary, noting the date, start time and end time of each session (in order to assess adherence to the sessions).
  Other Names: Period 1 - Booklet
  Arms: CONTROL
Other: Second period of the home-based adapted physical activity program with an exercise booklet. — Participants will receive a self-programme in the form of a booklet containing specific HIIT-type exercises adapted to their AIS. The programme is to be carried out at home over a 12-week period, with 3 45-minute sessions per week. The exercises are taken from the same database. Each participant in the CONTROL group will be encouraged to keep a follow-up diary, noting the date, start time and end time of each session (in order to assess adherence to the sessions).
  Other Names: Period 2

SUMMARY:
This study is a randomised controlled trial designed to compare two adapted physical activity treatments for adolescent idiopathic scoliosis (AIS). The main hypotheses it aims to address are as follows:

* Treatment with a HIIT (High-Intensity Interval Training) type training program via tele-rehabilitation, supervised by an adapted physical activity teacher, is effective in AIS.
* A 12-week physical activity program maintains this efficacy over the long term. To test this hypothesis, Two groups of adolescents will be evaluated: a first group made up of non-athletic adolescents suffering from Idiopathic Scoliosis who will benefit from a tele-rehabilitation (physical activity sessions at home supervised by a teacher in adapted physical activities by video). A second group, control, also made up of non-athletic adolescents suffering from Idiopathic Scoliosis who will benefit from a self-program at home consisting of exercises specific to their scoliosis.

DETAILED DESCRIPTION:
AIS is a deformity affecting 2% of adolescents between the ages of 10 and 16. It is a potentially severe condition with repercussions that impair the quality of life. Complications include respiratory issues (chronic restrictive insufficiency), pain and functional problems (chronic pain, evolving deformities even after growth cessation), bone-related concerns (osteopenia), psychological impacts (loss of self-esteem, tendency towards anxiety and depression), postural alterations (orthostatic postural control impairment), and aesthetic issues (deterioration of self-image).

The etiopathogenesis of AIS is not fully understood. Conventional treatments typically involve a combination of rehabilitation sessions and the use of a brace. Occasionally, corrective surgery (arthrodesis) may be necessary. There is a broad scientific consensus emphasizing the significant role of regular physical and sports activities (PSA) in AIS, as they improve its various comorbidities and complications.

Simultaneously, several epidemiological studies highlight insufficient engagement in PSA among adolescents, especially in France. This deficiency is more pronounced among girls, who are also eight times more affected by AIS than boys. Various factors contribute to adolescents' lack of interest in PSA, including excessive screen time, limited (geographical or economic) access to sports facilities, and a shortage of time and motivation.

Medical follow-up consultations for patients with AIS present an opportunity to underscore the importance of regularly engaging in PSA. It is also emphasized that these activities can be performed at home through specific self-programmed routines (adapted exercise booklets) provided to patients. Since the March 2020 covid-related lockdown, the investigators have observed that patients are making little use of the exercise books provided as part of their medical monitoring and are increasingly turning to online sports applications. This is an advantage as it allows adolescents to combine screen activities with PSA.

However, drawbacks include the non-specificity of the exercises offered, which may not always be suitable for AIS, and the lack of consistency over time, potential sources of inefficiency. Therefore, the aim to facilitate access to tailored PSA in a population of adolescents with AIS.

Various studies suggest that tele-rehabilitation is a credible therapeutic alternative applicable in key areas of pediatric rehabilitation. High-Intensity Interval Training (HIIT) programs, a method of PSA involving intervals of high intensity, are effective, particularly suitable for adolescents, and feasible through tele-rehabilitation.

The hypothesis is that an intervention involving a HIIT training program through tele-rehabilitation, supervised by an Adapted Physical Activity (APA) teacher, is effective in AIS.

To test this hypothesis, the investigators propose to compare the effectiveness of PSA at home over 12 weeks (PERIOD 1) in two groups of adolescents with AIS: a test group or TELE-APA group, which will receive an individualized, specific HIIT program tailored to each patient's scoliosis through tele-rehabilitation, supervised by an APA teacher, and a CONTROL group, which will receive a PSA program at home based on specific exercise booklets, of the HIIT type, adapted to each patient's scoliosis. After the third month, both groups will be followed for an additional 12 weeks (PERIOD 2), during which they will receive only a PSA program at home, in the form of an exercise booklet, of the HIIT type, adapted to each patient's scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* Affiliated to a social security system
* Having signed the consent after clear and fair information adapted to her age
* Obtained signed consent from at least 1 of the 2 parents or holders of parental authority, after clear and fair information
* Subject presenting an AIS defined by the existence of a three-dimensional deformity three-dimensional deformity of the spine associating a frontal deviation measured by by the frontal radiographic angle of Cobb which must be at least 15°, but less than 40°, and a vertebral rotation attested by the presence of a presence of at least 5° of gibbosity on Bunnel's scoliometer.
* Subject with front and side radiographs of the total spine, according to the EOS EOS technique, under load, less than 3 months old
* Risser test < 4/5 (EOS radiographs less than 3 months old)
* Subject not practicing any regular extracurricular physical activity (including regular (regular = at least 1 hour per week), for at least 6 months.
* Internet connection at home allowing tele-rehabilitation in a dedicated a dedicated room for the time of the session with a free surface of minimum 4m² on the floor, without any obstacle up to the ceiling.
* Compatibility with the technical requirements: access to a screen screen (computer or laptop, tablet...), with a minimum size of 8 inches (diagonal of 8 inches (diagonal of 20 cm), with an integrated or connected HD webcam connected, and a good quality sound, screen placed on a stable surface surface with a minimum height of 75cm and enough distance to see the to perceive from the camera the whole working area (4m²).

Exclusion Criteria: (One criterion is sufficient for non-inclusion)

* Subject with secondary scoliosis: neurological, orthopedic, malformative...
* Placement of a corset or rehabilitation for less than 3 months
* BMI ≤15 or ≥ 30
* Partial or total medical contraindication of any kind to the sports practice (examples: heart disease, unbalanced diabetes, juvenile polyarthritis, chronic painful joint pathology limiting physical performance, osteochondrosis of growth type Osgood-Schlater, Sever, Sinding-Larsen, osteochondritis, surgical sequelae limiting physical performance...)
* Inability to undergo the medical follow-up of the trial for psychological social or geographical reasons.

Ages: 13 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation to overall physical performance on an ergometer-rowing machine | Measured at the baseline and after 12 weeks
  Measurement of the time taken to complete 2000m as quickly as possible (in seconds)

SECONDARY OUTCOMES:
Evaluation of overall physical performance on an ergometer-rowing machine | Measured at 12 weeks and after 24 weeks
  Measurement of the time taken to complete 2000m as quickly as possible (in seconds)
Evaluation of perivertebral muscle performance (Plank) | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Maintaining maximum posture in seconds (s) in the Endurance plank test and two-side plank test.
Evaluation of perivertebral muscle performance (Rowing) | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Evaluation of maximum strength in kilograms (kg) in the Pull-down and seated row cable.
Indirect assessment of VO2 max | Measured at the baseline, after 12 weeks, and then after 24 weeks
  It will be evaluated from the Maximum Aerobic Speed (MAS), during the VAMEVAL test of Cazorla and Light on treadmill
The Ratings Perceveid Exertion for Children during exercise (RPE-C) | Measured at the baseline, after 12 weeks, and then after 24 weeks
  It will be carried out during the indirect evaluation of VO2 max, during the treadmill test, using the Borg scale adapted to treadmill test, using the Ratings Perceveid Exertion for Children (RPE-C). It is a pictorial, vertical scale graduated from 6 (low perception of effort) to 20 (maximum perception of effort). This evaluation will be requested every minute: the subject must indicate to the examiner (orally or by pointing) the score on the scale.
Assessment of motivation to change | Measured at the baseline, after 12 weeks, and then after 24 weeks
  It will be assessed by the questionnaire URICA (University of Rhode Island Change Assessment), composed of 32 statements, validated in children. The questionnaire allows us to determine in which stage the person is in his or her The URICA questionnaire makes it possible to determine in which stage the person is in his or her change: "Pre-contemplation", "Contemplation", "Determination", "Action".
Evaluation of attendance at adapted physical activity sessions | Once a week, up to 24 weeks
  It will be done by counting the number of physical activity sessions performed, either by the follow-up booklet (Control group for Control for Period 1, the 2 groups for Period 2), or by the count made by the the count made by the APA teacher who notes the presence of each patient each patient during the tele-rehabilitation sessions for the group TELE-APA group during Period 1.
Anthropometric evaluation (Height) | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Measurement of height in meters (m).
Anthropometric evaluation (weight) | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Measurement of weight in kilograms (kg).
Anthropometric evaluation (BMI) | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Weight and height will be combined to report BMI in kg/m^2)
Anthropometric evaluation by bioimpedance measurement | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Measurement of Lean Mass in kilograms (kg), Muscle Mass in kilograms (kg) and Fat Mass in kilograms (kg).
Analysis of the static vertical posture on a force platform SATEL® | Measured at the baseline, after 12 weeks, and then after 24 weeks
  The evaluation allows the analysis of the trajectory of the center of pressure, direct consequence of the body oscillations in standing position. The examination is carried out according to 3 modalities (eyes open on hard ground, eyes closed on closed on a hard floor, open eyes on a soft floor) allowing to obtain information on each sensory modality necessary for postural stabilization (visual, vestibular, and somesthesic related to the sole of the foot).
Evaluation of the EOS radiograph of the total spine in front (Type) | Measured at the baseline and then after 24 weeks
  Evaluation of the type of scoliosis according to Lenke's classification. Radiographic measurements in degrees of the Cobb angles, of the main curvature, of the thoracic kyphosis (between T4 and T12 and between T1 and T12), lumbar lordosis (between L1 and S1 and between L1 and L5).
Evaluation of the EOS radiograph of the total spine in front and in profile (Angle) | Measured at the baseline and then after 24 weeks
  Radiographic measurements in degrees of the Cobb angles, of the main curvature, of the thoracic kyphosis (between T4 and T12 and between T1 and T12), lumbar lordosis (between L1 and S1 and between L1 and L5).
Evaluation of the EOS radiograph of the total spine in front (Frontal deviation) | Measured at the baseline and then after 24 weeks
  Measurement in millimeters of the frontal spine deviation.
Evaluation of the EOS radiograph of the total spine in front (Risser) | Measured at the baseline and then after 24 weeks
  Evaluation of the Risser bone maturity test.
Photogrammetric morphostatic evaluation by surface topography | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Photogrammetric measurements in degrees of the Cobb angles, of the main curvature, of the thoracic kyphosis (between T4 and T12 and between T1 and T12), lumbar lordosis (between L1 and S1 and between L1 and L5).
  Measurement in millimeters of the frontal spine deviation.
Measurement of the main gibbosity | Measured at the baseline, after 12 weeks, and then after 24 weeks
  The gibbosity will be evaluated during the clinical examination, in degrees, using Bunnel's scoliometer, during the Forward Bending Test.
Assessment of quality of life by the Scoliosis Research Society (SRS) scale : SRS-18 | Measured at the baseline, after 12 weeks, and then after 24 weeks
  It is a specific scale for scoliosis, composed of 18 questions questions, classified into 5 themes (pain, function, body image, general satisfaction image, general satisfaction, treatment satisfaction). The global score score is between 18 (poor quality of life) and 90 (good quality of life). quality of life).
Satisfaction questionnaires | Measured at the baseline, after 12 weeks, and then after 24 weeks
  Satisfaction questionnaire at V2: the adapted physical activity teachers who supervised the tele-rehabilitation sessions, all the patients and a responsible representative fill in a satisfaction questionnaire at V2. A Visual Analogue Scale rated from 0 to 5 is used to assess the level of satisfaction with the treatment between V1 and V2 (Pleasure during the session, content of the sessions, safety of the sessions).
  - Additional question at V3: carried out only for the TELE-APA group. This is a double response question to define which adapted physical activity modality the patient preferred: tele-rehabilitation or self-programmed exercise book.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Catanzariti, Dr., Principal Investigator — Association des Paralysés de France
Locations (1):
- SMR Marc Sautelet, Villeneuve-d'Ascq, France

IPD SHARING:
Plan to Share IPD: No